CLINICAL TRIAL: NCT06572527
Title: The Effect of a Nurse-Led, Child Health Coordinated Physical Activity Program on Physical Activity Levels in Preschool Children: A Non-randomized Study
Brief Title: Child Health Coordinated Physical Activity Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Deniz Kocoglu-Tanyer, Professor Dr., Selcuk University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2023/75
Record Dates: First submitted 2024-07-27; First posted 2024-08-27 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Physical Activity; Children, Only; Nurse's Role; Body Weight Changes
MeSH Terms: conditions — Motor Activity; Body Weight Changes

STUDY DESIGN:
Intervention Model Description: Non-randomized, parallel assignment (1:1)
Who Masked: Outcomes Assessor
Masking Description: The outcomes obtained with the questionnaire form were collected from the families by the teachers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Nurse-Led Coordinated Physical Activity Program for Child Health, consisting of nurse, teacher, and family components was implemented by the researcher two days a week for six weeks. The interventions were last an average of 60 minutes each week. During this time, the nurse implemented a program, developed based on expert opinion and various guidelines, that directed students to be more active. Teachers were expected to encourage students and actively participate in the program. Families were regularly informed through the "family bulletin" and it was ensured that the program started at school was continued at home.
  Interventions: Behavioral: Physical Activity Program
- Control (No Intervention): No intervention was applied to the control group except for the regular physical activities they perform in their school life.

INTERVENTIONS:
Behavioral: Physical Activity Program — Nurse-Led Coordinated Physical Activity Program for Child Health," developed as part of the Coordinated Approach to Child Health program for preschool children.
  Arms: Intervention

SUMMARY:
This study was conducted as a non-randomized study to evaluate the effects of physical activity interventions developed with the Nurse-led Child Health Coordinated Physical Activity Program on the physical activity levels of preschool children.

Research hypotheses; H1a: The anthropometric measurements of the group receiving the intervention are different from the control group.

H1b: The physical activity levels of the group receiving intervention according to family reports are different from the control group

DETAILED DESCRIPTION:
The study group of the research consisted of 5-year-old students studying in kindergartens. The total number of students in kindergartens is 159 in the research area. Gpower 3.1.9.4 program was used to determine the sample size of the study. The sample size was determined as 42 ( 21 in the experimental and control groups) under a large effect size (0.80), an alpha value of 0.05 and a power level of 80%. It was decided to include a total of 52 students in the study by accepting a loss rate of approximately 20%.

Because it is known that it is important to promote physical activity at an early age, this study implemented interventions developed in accordance with the Coordinated Approach to Child Health Program, a program consisting of classroom, family, and student components. In the classroom component of the program, health education practices were prepared to teach children to identify, practice, and adapt physical activity habits to their lives through the classroom environment. In the family component of the program, there are interventions that ensure the participation of children, parents, and other family members to develop physical activity habits at home. Increasing physical activity in preschool children can be achieved by developing interventions that are fun and encourage children to be physically active in a structured classroom setting that promotes gross motor skills and moderate to vigorous physical activity during kindergarten and recess. In this study, a six-week program consisting of nurse, teacher, and family components developed in accordance with the Coordinated Approach to Child Health in Preschool Children program was implemented twice a week to evaluate its effects on physical activity in preschool children and its effectiveness in increasing physical activity.

The interventions averaged 60 minutes per week. Prior to implementation, school administrators and teachers were interviewed and informed about the purpose of the research and the implementation process. To inform parents and students about the research, the informed consent form and parent questionnaire were sent to parents in a sealed envelope and collected from students by teachers the next day. Informed consent was obtained by explaining the purpose and procedure of the study to the students whose parents had given their consent, and they were asked to complete the data collection instruments through the classroom teacher (pre-test). The post-test was administered 2 weeks after the completion of the study. The pre-test and post-test were administered by the teachers and the height-weight measurements were done by the nurse. No intervention was applied to the control group except for the physical activities they perform in their daily lives. Data collection instruments were administered to the control group in a similar manner and at the same time as the experimental group. The primary outcomes expected from the study are anthropometric measurements and physical activity levels. The research data was collected using the parent questionnaire developed by the researchers based on the literature and anthropometric measurements.

ELIGIBILITY:
Inclusion Criteria:

* Being 5 years old
* Being a student in kindergarten
* Volunteer for research
* Family consent to participate in the study
* The teacher of the class in which the student is enrolled agrees to participate in the study

Exclusion Criteria:

* Physical activity limitations due to medical conditions

  *After starting the study
* Absence from the program for at least two weeks
* If a situation arises during implementation that prevents participation in physical activity programs
* Withdrawal of consent.

Ages: 60 Months to 72 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 52 (Actual)
Dates: Start 2024-03-15 (Actual); Primary Completion 2024-05-20 (Actual); Study Completion 2024-06-05 (Actual)

PRIMARY OUTCOMES:
The parents' evaluation about their child's level of physical activity | Pre-intervention (T0) Two weeks after the end of the intervention (T1)
  This is a survey question. Parents rate their children's level of physical activity compared to their peers. (5-point scale from much more active to much less active)
The duration of watching TV or using a computer (in a day) | Pre-intervention (T0) Two weeks after the end of the intervention (T1)
  Time spent watching TV or using a computer
The status of organized planned physical activity | Pre-intervention (T0) Two weeks after the end of the intervention (T1)
  This question was developed based on the recommendation of at least 60 minutes of moderate-intensity physical activity per day. The status of moderate-intensity physical activity was explained with examples, and information about the child's activity status was obtained from the family for the past week . (Yes/no question) Expert opinion was obtained for the survey questions.
Time of playing outside | Pre-intervention (T0) Two weeks after the end of the intervention (T1)
  Time spent playing outside on weekdays and weekends,
The frequency of some activities | Pre-intervention (T0) Two weeks after the end of the intervention (T1)
  Number of activities per week (ranging from never to more than 3 times per week). This survey question is in accordance with the Department of Health and Human Services recommendation.
Anthropometric measurements | Pre-intervention (T0) Two weeks after the end of the intervention (T1)
  Change in body mass index, height and weight

CONTACTS AND LOCATIONS:
Locations (1):
- Emirdağ Fidan Ali Altıntaş Anaokulu, Afyonkarahisar, Turkey (Türkiye)